CLINICAL TRIAL: NCT04694833
Title: Self-assessment and Telerehabilitation Using Virtual Reality Devices and Serious Games to Improve Motor and Cognitive Impairments in Stroke Patients
Brief Title: Telerehabilitation Through Serious Games in Virtual Reality in a Stroke Population (AutoRReVi)
Acronym: AutoRReVi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROBIGAME; 1810108 (Other Grant/Funding Number: Région Wallonne - Economié Emploi Recherche - Win2Wal)
Record Dates: First submitted 2020-11-26; First posted 2021-01-05 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Hemiparesis; Cognitive Impairment; Healthy Subjects
MeSH Terms: conditions — Stroke; Paresis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Studies will be conducted in a single group of (a) stroke patients and (b) healthy subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke patients (Experimental): Stroke patients with hemiparesis and/or cognitive impairments (such as apraxia, aphasia and hemineglect)
  Interventions: Behavioral: Motor and cognitive virtual reality-based assessments; Behavioral: Motor and cognitive virtual reality-based serious games
- Healthy subjects (Experimental): Subjects who do not suffer from any pathology that could affect upper-limb motor function or cognition
  Interventions: Behavioral: Motor and cognitive virtual reality-based assessments; Behavioral: Motor and cognitive virtual reality-based serious games

INTERVENTIONS:
Behavioral: Motor and cognitive virtual reality-based assessments — Motor and cognitive testing in virtual reality
Behavioral: Motor and cognitive virtual reality-based serious games — Serious games implemented in virtual reality to rehabilitate motor and cognitive impairments.

SUMMARY:
After a stroke, individuals present with motor and/or cognitive impairments. These impairments limit activity, restrict participation and affect quality of life. Therefore, rehabilitation programs are provided from the earliest days. However, an important proportion of patients do not achieve the recommended amount of rehabilitation therapy (even in institutional systems). In fact, patients do not always have access to healthcare systems. Moreover, hospital resources and healthcare systems are often limited (especially in poor countries) which has led to the development of new cost-effective rehabilitation methods such as self-rehabilitation and tele-rehabilitation.

This study aims :

1. to develop and validate relevant self-assessments tools in virtual reality
2. to propose auto-adaptative virtual reality-based therapies based on the link between motor and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients (with hemiparesis or cognitive impairment such as apraxia, aphasia or hemineglect) OR healthy subjects
* Able to undersand simple instructions

Exclusion Criteria:

* Other disease that could affect upper limb motor function or cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Fugl-Meyer Assessment | Through study completion, on average 24 weeks
  Highly recommended scale that assess upper limb motor function (0% = worse outcome; 100% best outcome).
Box and Block Test | Through study completion, on average 24 weeks
  A measure of manual dexterity and activity that requires repeatedly moving 1-inch blocks from one side of a box to another in 60 seconds.
The Bells Test | Through study completion, on average 24 weeks
  A cancellation task, permits a quantitative and qualitative evaluation of visual neglect
Action Research Arm Test | Through study completion, on average 24 weeks
  A 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning). Items are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally).
System Usability Scale | Through study completion, on average 24 weeks
  Reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree

SECONDARY OUTCOMES:
Upper limb 3D position | Through study completion, on average 24 weeks
  Upper limb 3D position will be measured with different virtual reality devices (Oculus Quest, htc Vive, REAtouch). This will be done thanks to the headset's infra-red camera or the controller's inertial measurement units.
Upper limb peak velocity | Through study completion, on average 24 weeks
  Upper limb peak velocity will be measured with different virtual reality devices (Oculus Quest, htc Vive, REAtouch). This will be done by deriving 3D position (obtained previously thanks to the headset's infra-red camera or the controller's inertial measurement units) and extracting highest value.
Upper limb smoothness | Through study completion, on average 24 weeks
  Upper limb smoothness will be measured with different virtual reality devices (Oculus Quest, htc Vive, REAtouch). This will be done by deriving three times 3D position (obtained previously thanks to the headset's infra-red camera or the controller's inertial measurement units) and converting it to a logarithmic dimensionless jerk. Second option is to measure a spectral arc length (also computed from 3D position)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lejeune, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc - UCLouvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Woluwé, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorrentino G, Edwards MG, Baldini N, Mustile M, Lejeune T, Everard G. REAsmash-ET: a methodological framework for combined cognitive and motor assessment through eye-tracking and kinematic metrics in immersive VR search-and-reach task. J Neuroeng Rehabil. 2025 Dec 17. doi: 10.1186/s12984-025-01844-0. Online ahead of print. PMID 41408291
- [Derived] Everard G, Declerck L, Lejeune T, Edwards MG, Bogacki J, Reiprich C, Delvigne K, Legrain N, Batcho CS. A Self-Adaptive Serious Game to Improve Motor Learning Among Older Adults in Immersive Virtual Reality: Short-Term Longitudinal Pre-Post Study on Retention and Transfer. JMIR Aging. 2025 Mar 3;8:e64004. doi: 10.2196/64004. PMID 40053708
- [Derived] Ajana K, Everard G, Lejeune T, Edwards MG. An immersive virtual reality serious game set for the clinical assessment of spatial attention impairments: Effects of avatars on perspective? Technol Health Care. 2025 Jul;33(4):1626-1644. doi: 10.1177/09287329241296380. Epub 2025 Jan 17. PMID 39973878
- [Derived] Everard G, Burton Q, Van de Sype V, Bibentyo TN, Auvinet E, Edwards MG, Batcho CS, Lejeune T. Extended reality to assess post-stroke manual dexterity: contrasts between the classic box and block test, immersive virtual reality with controllers, with hand-tracking, and mixed-reality tests. J Neuroeng Rehabil. 2024 Mar 15;21(1):36. doi: 10.1186/s12984-024-01332-x. PMID 38491540
- [Derived] Burton Q, Lejeune T, Dehem S, Lebrun N, Ajana K, Edwards MG, Everard G. Performing a shortened version of the Action Research Arm Test in immersive virtual reality to assess post-stroke upper limb activity. J Neuroeng Rehabil. 2022 Dec 3;19(1):133. doi: 10.1186/s12984-022-01114-3. PMID 36463219
- [Derived] Everard G, Otmane-Tolba Y, Rosselli Z, Pellissier T, Ajana K, Dehem S, Auvinet E, Edwards MG, Lebleu J, Lejeune T. Concurrent validity of an immersive virtual reality version of the Box and Block Test to assess manual dexterity among patients with stroke. J Neuroeng Rehabil. 2022 Jan 22;19(1):7. doi: 10.1186/s12984-022-00981-0. PMID 35065678